CLINICAL TRIAL: NCT03796819
Title: Impact of Routine Lymphadenectomy on Prognosis of Patients Undergoing Curative Resection for Intrahepatic Cholangiocarcinoma
Brief Title: Routine Lymphadenectomy for Intrahepatic Cholangiocarcinoma
Acronym: LND for ICC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Ningxia Medical University (Other); Nanchang University (Other); Binzhou Medical University (Other); Shaanxi Provincial People's Hospital (Other); Shaanxi University of Chinese Medicine (Other); The Third Affiliated Hospital of Beijing University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XJTU1AFCRC2017SJ-007
Record Dates: First submitted 2019-01-06; First posted 2019-01-08 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2019-08

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: intrahepatic cholangiocarcinoma; surgery; lymphadenectomy; lymph node metastasis; prognosis
MeSH Terms: conditions — Cholangiocarcinoma; Lymphatic Metastasis | interventions — Lymph Node Excision

STUDY DESIGN:
Intervention Model Description: routine hepatoduodenal lymphadenectomy
Who Masked: Participant, Outcomes Assessor
Masking Description: patients would not be told about the lymphadenectomy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lymphadenectomy (Experimental): This group of patients would undergo routine hepatoduodenal lymphadenectomy combined with ICC resection
  Interventions: Procedure: lymphadenectomy
- No lymphadenectomy (No Intervention): This group of patients would not undergo hepatoduodenal lymphadenectomy when preoperative imaging and intraoperative exploration found no lymph node enlargement.

INTERVENTIONS:
Procedure: lymphadenectomy — Patients would undergo routine hepatoduodenal lymphadenectomy at the time of ICC resection
  Arms: lymphadenectomy

SUMMARY:
The role of routine lymphadenectomy (LND) in the surgical treatment of intrahepatic cholangiocarcinoma (ICC) remains controversial. The investigators' multi-institutional retrospective study have showed an increasing adoption of LND among patients undergoing curative resection for ICC during the last decade. The current prospective and randomized study based on a multi-institutional collaboration would investigate whether routine LND would benefit patients in short- and long-term survival remains.

DETAILED DESCRIPTION:
Intrahepatic cholangiocarcinoma (ICC) is the second most common primary liver cancer and its incidence is increasing worldwide.Resection of the primary ICC tumor site within the liver represents the best curative treatment option. However, the role of lymphadenectomy (LND) at the time of surgery remains controversial with some centers considering it standard while other surgeons perform LND only in select circumstances. The utilization of LND may not only vary among different institutions, but also by geographic region. Specifically, data from East and West centers have noted a variation in the utilization of LND ranging 27%-100%.While several case series from Asia have noted that most centers do not regularly perform LND,other data from the West suggest that LND may be becoming more routine. Despite the lack of consensus among surgeons, the American Joint Committee on Cancer (AJCC) Staging manual recommends that the nodal basin be staged. Disease-specific staging for ICC was first introduced in the 7th edition of the AJCC staging manual published in 2010. The newly updated 8th edition of the AJCC staging system now recommends that 6 lymph nodes be evaluated to stage a patient with ICC.

The previous multi-institutional retrospective study from the investigators have showed an increasing adoption of LND among patients undergoing curative resection for ICC during the last decade. The current prospective and randomized study based on a multi-institutional collaboration would investigate whether routine LND would benefit patients in short- and long-term survival remains.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with intrahepatic cholangiocarcinoma by imaging or biopsy
* The tumor is limited in the liver with no distant metastasis, and the primary disease is resectable
* Preoperative imaging (e.g. CT, MRI, PET-CT, etc.) and intraoperative exploration found no nodal swelling or enlargement

Exclusion Criteria:

* The primary disease is unresectable with or without distant metastasis
* The liver function or general condition of patients does not permit surgery
* Preoperative imaging (e.g. CT, MRI, PET-CT, etc.) and intraoperative exploration found obvious nodal swelling or enlargement, which indicates lymphadenectomy should be performed
* Patients aged below 18 or older than 65 would be excluded
* Pregnant women would not be enrolled

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
1-year recurrence rate | 1 year after surgery (up to 1 year)
  compare the 1-year recurrence rate of patients undergoing lymphadenectomy and those not undergoing lymphadenectomy
3-year recurrence rate | 3 years after surgery (up to 3 years)
  compare the 3-year recurrence rate of patients undergoing lymphadenectomy and those not undergoing lymphadenectomy

SECONDARY OUTCOMES:
Postoperative morbidity | From the date of surgery to stitches off (up to 1 month)
  investigate the postoperative morbidity, such as hepatic failure, postoperative bleeding, superficial and deep site infection between lymphadenectomy and no lymphadenectomy groups
1-year overall survival | 1 year after surgery (up to 1 year)
  compare the 1-year overall survival rate of patients undergoing lymphadenectomy and those not undergoing lymphadenectomy
3-year overall survival | 3 years after surgery (up to 3 years)
  compare the 3-year overall survival rate of patients undergoing lymphadenectomy and those not undergoing lymphadenectomy

CONTACTS AND LOCATIONS:
Overall Officials: Yi Lv, MD, PhD, Study Chair — First Affiliated Hospital Xi'an Jiaotong University; Xu-Feng Zhang, MD,PhD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China